CLINICAL TRIAL: NCT04272073
Title: A High-PRotein Mediterranean Diet and Resistance Exercise for Cardiac Rehabilitation: a Pilot Feasibility Study
Brief Title: A High-PRotein Mediterranean Diet and Resistance Exercise for Cardiac Rehabilitation
Acronym: PRiMER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Liverpool John Moores University (Other)
Collaborators: University of Chester (Other)
Responsible Party: Principal Investigator, Richie Kirwan, Post-graduate researcher, Liverpool John Moores University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 19LJMUSPONSOR0092; 256927 (Other: IRAS)
Record Dates: First submitted 2020-02-10; First posted 2020-02-17 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Cardiovascular Diseases; Sarcopenic Obesity
Keywords: sarcopenia; obesity; sarcopenic obesity; body composition; cardiac rehabilitation; cardiovascular disease; metabolic syndrome
MeSH Terms: conditions — Cardiovascular Diseases; Sarcopenia; Obesity; Metabolic Syndrome | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: A single-centre, cross-sectional analysis of the prevalence of SO in CR patients followed by a single-centre, 2x2 factorial, open label controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (Active Comparator): Participants will perform standard cardiac rehabilitation involving weekly (1-3 days) aerobic-focused exercise sessions in community gyms.
  Participants will have received guidance on weight management and healthy eating from cardiac rehabilitation staff but will not receive any further dietary support.
  Interventions: Other: Standard Dietary Advice; Other: Standard Cardiac Rehabilitation Exercise
- High-Protein mediterranean Diet and Resistance Exercise (Experimental): Participants will be asked to perform resistance exercise. This involves weights or weight machines aimed at building muscle strength. Participants will be required to attend 3 sessions per week and each session is expected to last approximately 45 minutes.
  Personalised dietary advice: we will ask participants to make changes to their diet to adapt it to a high-protein, Mediterranean-style diet
  * eating more fruit and vegetables,
  * reducing commercial pastries, and replacing refined carbohydrate foods (white bread, white rice, white pasta) by wholegrains (wholegrain bread, rice and pasta),
  * replacing butter and margarine by olive oil as the main culinary fat,
  * reducing fatty meat and replacing by lean meat, fish, and legumes (peas, beans, lentils), and by high-protein, low fat foods, such as low-fat dairy (participants will be provided with 2 dairy-based protein shakes to consume each day).
  Interventions: Other: High-Protein Mediterranean Diet; Other: Resistance Exercise

INTERVENTIONS:
Other: High-Protein Mediterranean Diet — As in arm/group descriptions
  Arms: High-Protein mediterranean Diet and Resistance Exercise
Other: Resistance Exercise — As in arm/group descriptions
  Arms: High-Protein mediterranean Diet and Resistance Exercise
Other: Standard Dietary Advice — As in arm/group descriptions
  Arms: Standard Care
Other: Standard Cardiac Rehabilitation Exercise — As in arm/group descriptions
  Arms: Standard Care

SUMMARY:
Cardiovascular disease is responsible for a quarter of all deaths in the UK and risk seems to be higher in cardiac rehabilitation (CR) with lower body weight which may be due to sarcopenci obesity (SO) or low muscle mass with high fat mass. The investigators aim to investigate the effect of a high protein Mediterranean diet and resistance exercise on improving lean mass and reducing risk markers of cardiovascular disease

DETAILED DESCRIPTION:
BACKGROUND Cardiovascular disease (CVD) in the UK is behind 1 in 4 deaths/year (>150,000 people), with coronary heart disease (CHD) being the most common type [1]. In addition to the loss of life, the economic cost of CVD is considerable; in 2015 healthcare for CVD alone in the UK amounted to £10.9 billion with a further £7.7 billion lost from the economy due to productivity loses [2].

Mortality figures due to CHD have been reduced recently, in part due to increased provision of cardiac rehabilitation (CR), a therapeutic approach based on exercise training to improve cardiac function, plus advice regarding smoking cessation, dietary changes and weight loss [3].

RATIONALE Most of the evidence on the benefit of CR examines the links between exercise and CV morbidity and mortality [4]; however, there is considerable evidence showing improvements in markers of cardiovascular risk through different dietary strategies [5]. Of particular relevance, results from studies on both the primary and secondary prevention of CVD suggest Mediterranean diet-based approaches are the most adequate to treat these patients [6-13].

Obesity, and in particular, visceral adiposity, is associated with cardiometabolic (CM) risk markers (e.g., high cholesterol and triglycerides levels, HbA1c, etc.) [14-16], however, an "obesity paradox" appears to exist in the cardiac population, where increased mortality has been linked to low body mass index (BMI) [17, 18]. However, low lean body mass (LBM) is the likely driver of this phenomenon due to sarcopenia, a progressive loss of LBM associated with aging [19]. Patients with a combination of low LBM and abdominal distribution of body fat, known as sarcopenic obesity (SO), are at greater risk of CVD, exacerbated in CR [20-23]. Thus, increasing relative LBM content, rather than simply promoting weight loss, may be an appropriate target in CR patients.

One particular barrier to maintaining or accruing LBM is the presence of anabolic resistance in older adults, which can result in a reduced muscle protein synthetic (MPS) response to both exercise and the ingestion of currently recommended intakes of protein [24]. Protein intakes above currently recommended levels (1.0-1.5 g/kg/BW) [25] combined with sufficiently intense resistance training [26] can overcome this anabolic resistance and positively influence muscle mass, ultimately leading to greater improvement in body composition, when accompanied by a reduction in total body fat mass [27].

RESEARCH QUESTION The investigators aim to determine the prevalence of sarcopenic obesity in a CR population and how this body composition relates to markers of cardiometabolic health. As there is no consensus definition of SO, multiple definitions, along with their relationship with CM risk markers, will be investigated.

The investigators aim to investigate to what extent a high-protein Mediterranean-style diet and resistance exercise, can augment LBM. Furthermore, the investigators will ascertain whether the above interventions improve markers of cardiometabolic health.

Therefore, the investigators will conduct a feasibility study with embedded pilot to obtain preliminary data on the practical and clinical considerations and cost-effectiveness of the proposed interventions, in preparation for an appropriately powered randomised controlled trial for increasing lean mass and improving cardiometabolic risk markers in patients with SO.

STUDY DESIGN AND METHODS OF DATA COLLECTION AND DATA ANALYSIS A single-centre, 2x2 factorial, non-randomised, open label controlled trial.

RANDOMISATION AND BLINDING All participants will be assigned to their group by self-selection of the desired intervention arm. Due to the nature of the intervention, blinding will not be possible.

INTERVENTIONS Approximately 40 patients will be asked to take part in the diet and exercise intervention, which will last 12 weeks. Participants at this stage will be allocated to one of two groups: 1) standard CR; 2) a high-protein, healthier diet plus resistance exercise.

Personalised dietary advice: if allocated to groups 2, the investigators will ask participants to make changes to their diet to adapt it to a high-protein, Mediterranean-style diet. Research shows that Mediterranean-style diets can reduce cardiovascular risk, and although there are different versions of this type of diet, they all have in common:

* eating more fruit and vegetables,
* reducing commercial pastries, and replacing refined carbohydrate foods (white bread, white rice, white pasta) by wholegrains (wholegrain bread, rice and pasta),
* replacing butter and margarine by olive oil as the main culinary fat,
* reducing fatty meat and replacing by lean meat, fish, and legumes (peas, beans, lentils), and by high-protein, low fat foods, such as low-fat dairy (participants will be provided with 2 high-protein dairy products to eat each day).

Participants will receive personalised guidance to help follow the new diet in the form of sessions at their community CR centre along with guide books and recipe guides. The goal is to make small, easy changes to their current eating habits, so the diet will be easy to follow. All foods included will be affordable and easy to find in local supermarkets (shopping guides will be provided), and the investigators will provide suggestions and recipes to prepare food. Participants will also receive dairy protein-based protein shakes and will be asked to consume these 2X per day, providing 25g of protein per serving for a total of 50g of supplemental protein per day.

If allocated to groups 1, participants will be asked to follow the diet recommendations given during phase 3 of CR.

Resistance exercise: if allocated to group 2, participants will be asked to perform resistance exercise. This involves weights or weight machines aimed at building muscle strength. Participants will be shown how to do the exercises by qualified instructors (BACPR cardiac rehabilitation certified) in the community centre where they carry out their current phase 3 cardiac rehabilitation. All exercises have been deemed safe for cardiac rehabilitation patients and an instructor will be available at all exercise sessions should they need assistance. Participants will be required to attend 3 sessions per week and each session is expected to last approximately 45 minutes.

If allocated to groups 1, participants will be asked to continue with the standard, aerobic-style exercise (treadmills, rowing machines, elliptical trainers) they have used in phase 3 of CR. This will also require 3 sessions per week.

SUBSEQUENT VISITS

All participants will have to attend two appointments at LJMU. The first visit will be just before beginning the intervention, and the second immediately after completing the intervention. Visits are expected to last 45-60 minutes and will entail:

BASELINE AND ENDPOINT ASSESSMENTS

To be carried out at LJMU Byrom St campus (L3 3AF) by the PhD student. The visit is expected to last 30 minutes and will entail:

i) Assessing body composition. This will be done in three different ways.

* Firstly, the investigators will measure participant height using a stadiometer and waist circumference using a tape measure.
* Secondly, the investigators will use a bioelectrical impedance analysis scale to measure lean body mass, total body fat mass and visceral fat mass.
* Thirdly, the investigators will perform a DXA (Dual-energy X-ray Absorptiometry) scan for 15-20 minutes which allows us to create an image of the distribution of lean body mass and fat mass.

ii) Taking blood pressure • Following standard protocol, participants will be asked to sit for 5 minutes before the investigators take blood pressure; the investigators will measure it three times to ensure an accurate reading.

iii) A venous blood sample

• The investigators will take about 8 teaspoons of blood. Particpants will need to fast for at least 12 hours prior to their appointment (although water is encouraged), as otherwise this may affect the result of the test.

iv) Food diaries (prior to lab appointments)

* Prior to second and third lab visits, participants will given a template of a three-day food diary, which they will need to complete the week before their lab appointment (on three working days plus one weekend or festive day, non-consecutive whenever possible), and bring with them on the morning of the visit. Participants will be contacted the day before to remind them of their appointment and what they must bring.

  (v) Mediterranean Diet Score
* Participants will fill in a brief 13-question questionnaire regarding the frequency of their intake of certain foods

(vi) Sarcopenia quality of life questionnaire • Participants will fill in a brief questionnaire regarding the current impact of sarcopenia on their quality of life

vii) Grip strength test

• Will be tested using a device that one squeezes as hard as possible (grip strength dynamometer). The investigators will do this three times to ensure an accurate reading.

STUDY SETTING This is a single centre study with all data collection taking place in LJMU, Byrom St. campus. All exercise will be carried out at the participants community CR centre, supervised by trained members of the community CR program.

STATISTICS AND ANALYSIS Cross-sectional study: from the results of body composition analysis, the prevalence of Pilot study: comparisons between intervention groups for all outcome measures will be performed by means of mixed model ANOVA, to account for inter-subject (differences between treatments) and intra-subject (differences between baseline and endpoint) variability. Since a sample size calculation will not be conducted for this component, interpretation of the results will be largely descriptive and focused on confidence limits around parameter estimates.

Statistical significance will be set at p<0.05, and all analyses will be conducted using IBM SPSS Statistics v25 (SPSS Inc., Chicago, IL).

PARTICIPANT RECRUITMENT STUDY PARTICIPANTS Participants will be recruited from Liverpool Heart & Chest Hospital Cardiac Rehabilitation unit. Participants in the intervention trial will have recently completed phase 3 CR, will have been deemed as cardiac stable, and will be willing to participate in phase 4 CR (Activity for Life). The minimum age restriction for participants will be 40-years

The sample size for the feasibility study has been arbitrarily kept small (20 participants per intervention group) to allow ease of recruitment and management of participants before development into a fully powered randomised controlled trial.

RECRUITMENT TECHNIQUE Participants will be approached by members of their clinical care team at LHCH, who will invite them to participate and confirm they are willing to be contacted by the research team for more information. Please refer to 6.5 for further details.

PARTICIPANT IDENTIFICATION Eligible participants will be recruited from patients recently referred to cardiac rehabilitation (Liverpool Heart & Chest Hospital Cardiac Rehabilitation Unit), which is where the investigators will start the study. In collaboration with the LHCH Cardiac Rehabilitation Unit, eligible participants will first be identified by the clinical care team.

Eligible participants will be approached by members of the Knowsley Community Cardiovascular Services team, part of Liverpool Heart & Chest Hospital Cardiac Rehabilitation unit. Participants will be informed of the research and provided with a participation information sheet and asked to reply with their interest after 24 hours. They will then be contacted by the PhD student.

SCREENING AND ELIGIBILITY ASSESSMENT Initial screening will be carried out via initial phone conversation with potential participants referred via the CR team at LHCH.

INFORMED CONSENT The participant must personally sign and date the latest approved version of the Informed Consent form before any study specific procedures are performed.

Written and verbal versions of the Participant Information and Informed Consent will be presented to the participants detailing no less than: the exact nature of the study; what it will involve for the participant; the implications and constraints of the protocol; the known side effects and any risks involved in taking part. It will be clearly stated that the participant is free to withdraw from the study at any time for any reason without prejudice to future care, without affecting their legal rights, and with no obligation to give the reason for withdrawal.

The participant will be allowed as much time as wished to consider the information, and the opportunity to question the Investigator, their GP or other independent parties to decide whether they will participate in the study. Written Informed Consent will then be obtained by means of participant dated signature and dated signature of the person who presented and obtained the Informed Consent. The person who obtained the consent must be suitably qualified and experienced, and have been authorised to do so by the Chief/Principal Investigator. A copy of the signed Informed Consent will be given to the participant. The original signed form will be retained at the study site.

DISCONTINUATION/WITHDRAWAL OF PARTICIPANTS FROM STUDY

Each participant has the right to withdraw from the study at any time. In addition, the Investigator may discontinue a participant from the study at any time if the Investigator considers it necessary for any reason including:

* Pregnancy
* Ineligibility (either arising during the study or retrospectively having been overlooked at screening)
* Significant protocol deviation
* Significant non-compliance with treatment regimen or study requirements
* Withdrawal of Consent
* Loss to follow up

Should a participant wish to withdraw from the study, their anonymised data will be retained for 10 years. Their data may still be included in the analysis if they withdraw after completing the intervention, and for reasons that do not affect the study outcomes. If the participant wants their data to be removed from the study, they may contact us and request such.

Withdrawn participants may be replaced should sufficient time and resources be available.

The reason for withdrawal by researcher (and by participant, if this information is volunteered) will be recorded in a study file.

DATA MANAGEMENT ACCESS TO DATA Direct access will be granted to the research team, authorised representatives from the Sponsor and host institution for monitoring and/or audit of the study to ensure compliance with regulations.

DATA RECORDING AND RECORD KEEPING The information provided as part of the study will be anonymised. The investigators will use codes to label, trace and identify samples, records and questionnaires; the investigators will never use any personal data from which participants can be identified, such as name, initials, or date of birth.

Documents that include personal data (such as the consent form, or contact details) will be stored on password-protected computers and locked filing cabinets at LJMU, accessed only by the research team. They will be destroyed upon completion of the study, unless they would like a copy of the final study results; in that case, the investigators will retain their names, phone numbers and email addresses, so the investigators can contact them later. The results should be available approximately 1 year after the study is completed; participant personal data will be then deleted.

Research data will be stored in databases using the codes as identifiers, never personal data, and they will be kept in password-protected computers only accessed by the research team. Samples will be booked into a database and receive a laboratory code, with only those involved in the research having access. All data and samples will be destroyed after 10 years.

The names of participants will never be published in any communication of results and findings.

SAMPLE HANDLING

Blood samples will be processed and stored according to current UK regulations and rules of good research practice (Human Tissue Act 2004), and will be kept for a maximum of 10 years. Briefly, blood samples will be processed immediately after collection, and the serum will be stored in a secure freezer in the Life Sciences Building at LJMU's Byrom St campus. All samples will be stored pseudo-anonymously; this means that all identifiable information will be removed and replaced by a code to allow the research team to trace the samples and match them with the other measurements (body weight, muscle mass measures, etc.). Once all participants have completed the intervention, samples will be analysed. Once the specified storage period ends, all samples will be disposed of following current UK regulations.

ETHICAL AND REGULATORY CONSIDERATIONS DECLARATION OF HELSINKI The Investigator will ensure that this study is conducted in accordance with the principles of the Declaration of Helsinki and relevant regulations

ASSESSMENT AND MANAGEMENT OF RISK Participants will be scanned by a DXA scanner, which will involve use of small doses of ionising radiation, though this is a minimal amount compared to other medical imaging techniques, such as standard X-ray and CT scans. The DXA scan would be equal to approximately 2 microsieverts (μSv); this is compared to 20 microsieverts for a chest X-ray and 10,000 microsieverts for a CT scan. It is also less than a transcontinental flight (40 μSv) and one day of natural background radiation (8 μSv).

Great care will be taken to ensure vulnerable people (for example, pregnant women) will not be permitted to take part, both during the initial screening and recruitment, and also during the scans where mandatory exclusion criteria are checked before the scan can begin.

The study will limit the involvement of each participant to three scans, and they will be fully informed as to the exposure they will have, should they choose to participate. The radiation exposure is so low that no shielding of the room or of the person conducting the scans is necessary; therefore, the anticipated risk to the participant is negligible.

The participants are being asked to be involved in a study which has a central focus on body weight and composition, which can be a very sensitive subject. As the participants will be willing volunteers for the study, it is expected that only people who are comfortable with this issue will be involved. Additionally, the participants can request for their bio-impedance and anthropometric measurements to be taken by a member of the research team of the same gender. They can also request a chaperone to be present during the procedure. Privacy and confidentially will be ensured when taking measurements, and all data will be anonymised upon collection and storage.

In addition, participants will be reminded that they can withdraw and remove themselves from the situation (and the study) at any time.

For the DXA scans, questionnaires and anthropometric measurements, it is not anticipated that there will be significant inconvenience for those who choose to take part in this project, as their time involvement is minimal at 45 minutes per visit, and the investigators will do their best to accommodate their visit times to their preferences and availability (within the limits of the research requirements).

Participants will be made aware of the requirements of the dietary intervention while seeking consent, and it is expected that those who are comfortable with this dietary change will be involved. The dietary intervention will not use difficult to source ingredients and will be tailored to suit the tastes of the participants. Various recipes and food substitutions will be provided to participants at the beginning of the protocol. The high-protein diet of the protocol would only be potentially detrimental to individuals who have renal deficiency, and therefore this is one of the studies exclusion criteria. Participants will also receive regular contact from the PhD student regarding their adherence.

Participants will be made aware of the requirements of the exercise intervention while seeking consent, and it is expected that those who are comfortable with this change in physical activity will be involved. All participants will have received exercise tolerance tests as part of their NHS cardiac rehabilitation and will be cleared for the exercise protocol. They will also receive instruction from a collaborator suitably trained in exercise for cardiac rehabilitation regarding how to safely complete the exercise protocol.

The involvement of the participants and their data will be kept confidential, with no personal identifying data being present on questionnaires, forms or DXA scans. The unique code that can identify a participant will be kept on a secure system that can only be accessed by the research team. Therefore it is not expected that there will be a significant risk of a confidentiality breach.

Should the participant disclose information indicating a risk of potential harm to themselves or others, the appropriate authority will be contacted (LHCH, patient's GP, police etc,).

PARTICIPANT CONFIDENTIALITY The data custodian will be the PhD student. All investigators and study site staff must comply with the requirements of data protection legislation with regards to the collection, storage, processing and disclosure of personal information and will uphold the Act's core principles.

Information provided as part of the study will be anonymised. The investigators will use codes to label, trace and identify samples, records and questionnaires; the investigators will never use any personal data from which participants can be identified, such as name, initials, or date of birth.

Documents that include personal data (such as the consent form, or contact details) will be stored on password-protected computers and locked filing cabinets at LJMU, accessed only by the research team. They will be destroyed upon completion of the study, unless participants would like a copy of the final study results; in that case, the investigators will retain their name, phone number and email address, so the investigators can contact them later. Their personal data will then be deleted

Research data will be stored in databases using the codes as identifiers, never personal data, and they will be kept in password-protected computers only accessed by the research team. Samples will be booked into a database and receive a laboratory code, with only those involved in the research having access. All data and samples will be destroyed after 10 years.

The names of participants will never be published in any communication of results and findings.

EXPENSES AND BENEFITS Participants will not be reimbursed for travel expenses incurred while participating in the study

Participants in the high protein diet groups will be provided with 2 high-protein yoghurts per day for the duration of the trial.

The diet and exercise chosen in this study have been shown to have a number of benefits:

* High-protein foods may increase satiety after a meal, reducing hunger.
* This may also lead to a lower calorie intake and consequential potential weight loss.
* This may lead to a loss of fat mass, improving body composition.
* Muscles may grow and become stronger, meaning everyday activities will feel easier.
* Blood sugar levels may improve due to healthier muscles helping with blood sugar control.
* Blood cholesterol and fats may improve, reducing risk of further cardiac events.

OTHER ETHICAL CONSIDERATIONS In the unlikely event of finding any abnormalities or anything of clinical significance, the findings will be checked by a clinical specialist. If the specialist feels that the abnormality was medically important, they will discuss the implications with the participant and arrange for further investigations as necessary. Participants will not be informed unless the doctor considers the finding has clear implications for their current or future health. It is important to note that data collected are not carried out for diagnostic purposes, and therefore the data are not a substitute for a clinical appointment. Rather, the data are intended for research purposes only.

RESEARCH ETHICS COMMITTEE (REC) AND OTHER REGULATORY REVIEW & REPORTS

* Before the start of the study, a favourable opinion will be sought from from the UK Health Departments Research Ethics Service NHS REC for the study protocol, informed consent forms and other relevant documents e.g. advertisements
* Approval will be obtained from LJMU REG (and Co-Sponsors) for any amendments to, or changes of status in the study prior to submission to the REC that ethically approved the study and any other regulatory authorities
* All correspondence will be retained.
* The protocol, informed consent form, participant information sheet and any proposed advertising material will be submitted to the HRA for written approval.
* Annual Progress Reports will be submitted to the NHS REC which gave the favourable opinion, the HRA (hra.approval@nhs.net) and the Sponsor (Sponsor@ljmu.ac.uk) on the anniversary of NHS REC Favourable Opinion, and annually thereafter until the End of Study Declaration has been submitted to the NHS REC which gave the favourable opinion, the HRA and the Sponsor
* Upon the completion of the study an End of Study Declaration (within 90 days of the end of the study) and End of Study Report (within 12 months of the end of the study) will be submitted to the NHS REC which gave the favourable opinion and LJMU REG (sponsor@ljmu.ac.uk)
* Annual Progress Reports will be submitted to the NHS REC which gave the favourable opinion and the Sponsor (Sponsor@ljmu.ac.uk) on the anniversary of HRA approval, and annually thereafter until the End of Study Declaration has been submitted to the NHS REC which gave the favourable opinion and the Sponsor.
* Upon the completion of the study an End of Study Declaration (within 90 days of the end of the study) and End of Study Report (within 12 months of the end of the study) will be submitted to the NHS REC which gave the favourable opinion and LJMU REG (sponsor@ljmu.ac.uk)
* Early termination or suspension of the research will be reported to all relevant review bodies and the Sponsor (sponsor@ljmu.ac.uk) within 15 days.

SCIENTIFIC REVIEW

The study protocol went through successive stages of scientific review:

1. It was first reviewed and approved for support under the cross-faculty PhD funding scheme. The panel reviewing the proposals was formed by staff from the Faculty of Science, Faculty of Education, Health and Community, and the Institute of Health Research, LJMU.
2. The study was subsequently reviewed and approved by the Service Users Research Endeavour (SURE) Group of the Liverpool Heart and Chest Hospital.
3. Finally, our study protocol was presented at and approved by the Research and Innovation Committee of the Liverpool Heart and Chest Hospital.

All different stages of review were carried out by independent reviewers, both internal (from LJMU) and external (LHCH), meeting the requirements of Level 4 studies.

PROTOCOL COMPLIANCE Protocol adherence will be monitored with weekly phone call with each participant, carried out by the PhD student. This will also be an opportunity for participant to inform the PhD student of any adverse events they have experienced.

Accidental protocol deviations can happen at any time. They will be adequately documented on the relevant forms and reported to the Chief Investigator and Sponsor immediately.

Deviations from the protocol which are found to frequently recur are not acceptable, will require immediate action and could potentially be classified as a serious breach.

The Investigator may discontinue a participant from the study at any time if the Investigator considers it necessary for any reason. Such occurrences will be detailed in the individual participant study logs

CONTRACTS AND AGREEMENTS A standard Non-Commercial Model Agreement (mNCA) will be negotiated with Liverpool Heart & Chest Hospital

A research passport (letter of access) will be applied for, for the PhD student who will undertake the research within the NHS.

DEFINITION OF END OF STUDY The end of study is the date of completion of analysis of samples.

END OF STUDY AND ARCHIVING The end of study is the date of the last visit of the last participant. Relevant consent forms will be obtained for each participant, allowing for the samples to be stored and data to be archived for at least 10 years.

ACCESS TO THE FINAL STUDY DATASET Aim: to describe who will have access to the final dataset The PhD student, all supervisors and the lead clinician will have access to the full dataset. The study will allow site investigators to access the full dataset if a formal request describing their plans is approved by the steering group. Any secondary analysis will only be undertaken with the consent of the participants. All patient documentation will reflect the future use of data in research.

ELIGIBILITY:
Stage 1:

Inclusion Criteria:

* Informed consent given
* Referral to cardiac rehabilitation program
* Ability to attend screening at Liverpool John Moores University

Stage 2:

* Informed consent given
* Meeting selected criteria to define sarcopenic obesity (dependent on analysis from stage 1)
* Ability to attend screening at Liverpool John Moores University
* Cardiac function deemed stable after phase 3 cardiac rehabilitation

Exclusion Criteria:

* Inability to perform resistance exercise (determined by primary care team)
* Renal dysfunction
* Inability/unwillingness to digest/consume dairy products
* Admission to CR due to congenital or drug/alcohol-abuse induced cardiac events
* Pregnancy

Ages: 30 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2022-05-09 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Feasability of recruitment | 10 months
  Recruitment numbers over time course of study
Follow up rates | 18 months
  Number of participants that respond to follow up questionnaires
Acceptability of dietary intervention | 18 months
  Qualitative data from focus groups
Acceptability of exercise intervention | 18 months
  Qualitative data from focus groups
Adherence to exercise protocol | 12 weeks
  Number of exercise sessions actually attended out of number of prescribed sessions

SECONDARY OUTCOMES:
Change in appendicular skeletal muscle mass (DXA) | 12 weeks
  Appendicular skeletal muscle mass in kg as measured by DXA
Change in muscle mass (DXA) | 12 weeks
  Muslce mass in kg as measured by DXA
Change in muscle mass (BIA) | 12 weeks
  Muscle mass in kg as measured by SECA BIA monitor
Change in fat mass (BIA) | 12 weeks
  Fat mass in kg as measured by SECA BIA monitor
Change in visceral fat mass (DXA) | 12 weeks
  Visceral fat mass in kg as measured by DXA
Change in waist circumference | 12 weeks
  Waist circumference in cm as measured by anthropometric tape
Change in body weight | 12 weeks
  Body weight in kg as measured by scales
Height | 12 weeks
  Height in cm as measured by stadiometer
Change in waist:height ratio | 12 weeks
  Waist circumference in cm : height in cm
Improvement in cardiometabolic risk markers | 12 weeks
  Changes in cardiometabolic risk markers (e.g. lipid profile, fasting glucose, HbA1c etc).
Change in total cholesterol | 12 weeks
  Cholesterol in mmol/L
Change in HDL cholesterol | 12 weeks
  HDL cholesterol in mmol/L
Change in non-HDL cholesterol | 12 weeks
  non- HDL cholesterol in mmol/L
Change in fasting triglycerides | 12 weeks
  Fasting triglycerides in mmol/L
Change in fasting glucose | 12 weeks
  Fasting glucose in mmol/L
Change in Total cholesterol : HDL cholesterol ratio | 12 weeks
  Total HDL cholesterol in mmol/L : HDL cholesterol in mmol/L
Change in HbA1c | 12 weeks
  HbA1c in mmol/mol
Change in blood pressure | 12 weeks
  Blood pressure measured in mm/Hg
Change in grip strength | 12 weeks
  Grip strength measured in kg using grip strength dynamometer
Change in back/leg strength | 12 weeks
  Back/leg strength measured in kg using back/leg strength dynamometer
Change in mediterranean diet score | 12 weeks
  MEDAS questionnaire score in points out of 14
Change in sarcopenia Quality of life score | 12 weeks
  Sar-Q questionnaire score in points

CONTACTS AND LOCATIONS:
Overall Officials: Fatima Perez de Heredia Benedicte, PhD, Principal Investigator — Liverpool John Moores University
Locations (1):
- Knowsley Community Cardiovascular Services, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] McCullough D, Kirwan R, Butler T, Perez de Heredia F, Thijssen D, Lip GYH, Mills J, Davies IG. Feasibility of a high-PRotein Mediterranean-style diet and resistance Exercise in cardiac Rehabilitation patients with sarcopenic obesity (PRiMER): Study protocol for a randomised control trial. Clin Nutr ESPEN. 2021 Oct;45:492-498. doi: 10.1016/j.clnesp.2021.08.001. Epub 2021 Aug 15. PMID 34620360

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-01-06): https://cdn.clinicaltrials.gov/large-docs/73/NCT04272073/Prot_SAP_000.pdf
  • Informed Consent Form (2020-01-06): https://cdn.clinicaltrials.gov/large-docs/73/NCT04272073/ICF_001.pdf